CLINICAL TRIAL: NCT04434690
Title: Radiologic Results of One-Stage Bilateral TKR - One Surgeon Sequential vs. Two Surgeon Simultaneous: A Randomized Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Orkhan Aliyev, MD, Resident Doctor in Orthopaedic Surgery, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 71306642-050.01.04
Record Dates: First submitted 2020-06-13; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Gonarthrosis; Primary
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simultaneous (Experimental): 2 surgeons will perform simultaneous total knee arthroplasty in this group.
  Interventions: Procedure: Simultaneous bilateral total knee arthroplasty
- Single surgeon bilateral TKA group (Active Comparator): One surgeon will perform sequentially tptal knee arthroplasty in this group
  Interventions: Procedure: Sequenced bilateral TKA

INTERVENTIONS:
Procedure: Simultaneous bilateral total knee arthroplasty — Two surgeons bilateral TKA group
  Arms: Simultaneous
Procedure: Sequenced bilateral TKA — Single surgeon bilateral TKA group
  Arms: Single surgeon bilateral TKA group

SUMMARY:
Many surgeons and patients prefer bilateral total knee arthroplasty (TKA) under one anesthesia as single-stage administration. A single-stage bilateral TKA can be performed in two different ways: single-stage, two-team simultaneous bilateral TKA (two surgeons bilateral TKA), and single-stage, a sequential bilateral TKA (single surgeon bilateral TKA). The purpose of this study is to evaluate the radiological results in the single-stage bilateral TKA in terms of two surgeons bilateral TKA and single surgeon bilateral TKA.

DETAILED DESCRIPTION:
Investigators will enroll 136 participants with primary bilateral symptomatic knee osteoarthritis that will refractory to conservative treatment who will undergo bilateral TKA under single anaesthesia after 15.06.2020. Investigators will include patients who were less than 75 years old, with no history of malignancy, without severe extra-articular deformities, and without the systemic inflammatory disease, severe cardiac insufficiency, and morbid obesity (>40 kg/m2 or 35 or more and experiencing obesity-related health conditions). An informed consent form will be obtained from all patients.

ELIGIBILITY:
Inclusion Criteria:

Primary bilateral knee osteoarthritis with refractory to conservative treatment Patients who accept participation in the research and the randomization

Exclusion Criteria:

no history of malignancy less than 75 years old without severe extra-articular deformities severe cardiac insufficiency and morbid obesity without systemic inflammatory diseases

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Radiological examination | 14days
  Coronal and Sagittal Alignment

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No